CLINICAL TRIAL: NCT01390155
Title: Characterization of Ischemia Related Changes in Esophageal Electrocardiography
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Vogel Rolf, Prof. Dr. med., University Hospital Bern
Other Study IDs: 058/11
Record Dates: First submitted 2011-07-01; First posted 2011-07-08 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Artery Disease
Keywords: Electrocardiography; Coronary Artery Disease; Atrial Fibrillation; Heart Atria; Coronary Circulation; Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation; Ischemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Patients undergoing temporary myocardial ischemia produced by a one-minute balloon occlusion of the proximal left anterior descending coronary artery.
  Interventions: Procedure: Measurement of coronary collateral flow index
- 2: Patients undergoing temporary myocardial ischemia produced by a one-minute balloon occlusion of the proximal left circumflex artery.
  Interventions: Procedure: Measurement of coronary collateral flow index
- 3: Patients undergoing temporary myocardial ischemia produced by a one-minute occlusion of the proximal right coronary artery.
  Interventions: Procedure: Measurement of coronary collateral flow index
- 4: Patients undergoing temporary myocardial ischemia produced by a one-minute occlusion of the target vessel.
  Interventions: Procedure: Measurement of coronary collateral flow index

INTERVENTIONS:
Procedure: Measurement of coronary collateral flow index — One-minute balloon occlusion of the proximal left anterior descending coronary artery inducing a controlled short-time ischemic condition of a part of the myocardium and simultaneous evaluation of collateral flow.
  Groups: 1
Procedure: Measurement of coronary collateral flow index — One-minute balloon occlusion of the proximal left circumflex artery inducing a controlled short-time ischemic condition of a part of the myocardium and simultaneous evaluation of collateral flow.
  Groups: 2
Procedure: Measurement of coronary collateral flow index — One-minute balloon occlusion of the proximal right coronary artery inducing a controlled short-time ischemic condition of a part of the myocardium and simultaneous evaluation of collateral flow.
  Groups: 3
Procedure: Measurement of coronary collateral flow index — One-minute balloon occlusion of the target vessel (the vessel which shows a significant stenosis and accordingly requires a therapeutical intervention by balloon angioplasty and stenting) inducing a controlled short-time ischemic condition of a part of the myocardium and simultaneous evaluation of collateral flow.
  Groups: 4

SUMMARY:
Esophageal electrocardiography (eECG) has important advantages compared to standard ECG recordings.

Coronary artery disease leading to myocardial ischemia is very common and has potentially severe consequences for patients. To date, the investigators don't know the influence of ischemia on the eECG. The goal of the present study is to assess ischemic changes of the eECG induced by balloon occlusion of coronary arteries in patients undergoing coronary angiography.

DETAILED DESCRIPTION:
Background

Heart rhythm disorders frequently occur in the general population and potentially have serious consequences. Atrial fibrillation, the most common atrial arrhythmia, can lead to intracardiac blood clot formation an subsequent embolisation. Esophageal electrocardiography (eECG) provides detailed information about the electrical activity of the atria. Due to the good signal quality, eECG is a promising technique for rhythm monitoring.

Patients undergoing rhythm monitoring may also show signs of other cardiac diseases, particularly coronary artery disease (CAD) due to its high prevalence. It is therefore mandatory to define the ischemic changes in the esophageal ECG.

In CAD atherosclerotic processes narrow the lumen of coronary arteries and may cause exercise-induced ischemia (stable CAD). More importantly, there is also the risk of plaque rupture and subsequent blood clot formation. This cascade can lead to total occlusion of the coronary vessel and myocardial infarction.

Coronary angiography is used to determine the severity of coronary artery stenosis. This simple approach turned out to be useful in clinical routine. However, presence or absence of coronary collaterals is one of the reasons why coronary angiography alone may fail to define the clinical relevance of CAD. Collateral vessels as natural bypasses can grow and act as "backup" blood supply of the myocardial area at risk and can therefore reduce infarct size. The coronary wedge-pressure method is recognized as the scientific and clinical gold standard. Collateralization is an important confounder which also can "mask" ischemic changes on the ECG.

The surface ECG of an important portion of patients undergoing arrhythmia screening also shows signs of myocardial ischemia due to CAD or left ventricular hypertrophy. As with the surface ECG, it is conceivable that ischemic changes occur in the eECG. The characterization of ischemia related changes in eECG is crucial in order to guarantee the proper classification of eECG events. To date, the characterization of such changes is not adequate in order to allow the reliable clinical interpretation of eECG changes.

Objective

* To characterize changes in the esophageal ECG induced by myocardial ischemia due to short-time coronary occlusion.
* To determine the influence of coronary collateral vessels on these changes.

Methods

Patients referred for elective coronary angiography will be randomized to four groups:

1. Patients undergoing temporary myocardial ischemia produced by a one-minute balloon occlusion of the proximal left anterior descending (LAD) coronary artery.
2. Patients undergoing temporary myocardial ischemia produced by a one-minute balloon occlusion of the proximal left circumflex artery.
3. Patients undergoing temporary myocardial ischemia produced by a one-minute balloon occlusion of the proximal right coronary artery.
4. Patients undergoing temporary ischemia produced by a one-minute occlusion of the target vessel (the vessel which shows a significant stenosis and accordingly requires a therapeutical intervention).

During the occlusion, collateral flow indexes will be calculated. Simultaneously, surface ECG, esophageal ECG and intracoronary ECG will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for elective coronary angiography
* Age >/= 18 years
* Written informed consent to participate to this study

Exclusion Criteria

* Seve mitral- or aortic valve disease
* Acute coronary infarction
* Known bleeding diathesis
* Systolic blood pressure >200mmHg
* History of operations of the esophagus
* Active disease of the upper respiratory and gastroesophageal tract
* Radiofrequency ablation of atrial fibrillation, less than six weeks ago
* Right and left bundle branch block
* Significant Q-waves in the surface leads as indicators for prior myocardial infarction
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for elective coronary angiography due to suspected or known coronary artery disease.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
ST-segment-elevation/depression in the ECG at J-point and 80ms later | 0, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110 and 120 seconds after start of vessel occlusion

SECONDARY OUTCOMES:
Increase/decrease of T-wave amplitude | 0, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110 and 120 seconds after start of vessel occlusion
Relative ST-segment-elevation/depression | 0, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110 and 120 seconds after start of vessel occlusion
Sensitivity and specificity of the esophageal electrocardiogram detecting ischemic conditions (using the intracoronary ecg as gold standard) | at the end of occlusion, expected on average to be 60 seconds
New U-wave | during the whole occlusion time, expected on average to be 60 seconds
beat-to-beat alternans of the ST-segment | during the whole occlusion time, expected on average to be 60 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Vogel, MD, MD-PhD, Study Director
Locations (1):
- Dep. of Cardiology, Bern University Hospital, Bern, Canton of Bern, Switzerland